CLINICAL TRIAL: NCT00499629
Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of FXR-450 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety of FXR-450 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3213A1-1000
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Arm 1: FXR 450
  Interventions: Drug: FXR 450
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: FXR 450 — capsule, single oral doses from 10 mg to 450 mg
  Arms: 1
Drug: placebo — capsule similar to active drug
  Arms: 2

SUMMARY:
The primary purpose of the study is to evaluate the safety of FXR-450 in healthy subjects. This study will also evaluate pharmacokinetics (PK) of FXR-450 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential (WONCBP) aged 18 to 50 years inclusive at screening.
* Healthy as determined by the investigator on the basis of screening evaluations.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Exclusion Criteria:

* Any significant medical disease.
* History of cholecystectomy (removal of gallbladder).
* Any clinically important finding in physical examination, vital signs, 12-lead electrocardiograms (ECGs), or clinical laboratory test results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability | 4 days

SECONDARY OUTCOMES:
pharmacokinetics | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Facility, Philadelphia, Pennsylvania, United States